CLINICAL TRIAL: NCT04043767
Title: Prognostic Factors for Difficult Intubation in Pediatric Patients
Brief Title: Prognostic Factors for Difficult Intubation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Ngamjit Pattaravit, Primary investigator, Prince of Songkla University
Other Study IDs: difficult airway
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: The Predictors of Difficult Intubation in Pediatric Patients
Keywords: predictors, difficult intubation, pediatric patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients aged between 1-8 years: Pediatric patients aged between 1-8 years who scheduled for general anesthesia in elective surgery. Additional physical examinations which were including thyromental distances, hyomental distances and neck circumferences, was performed at one day prior surgery. Intubation was done by general anesthesiologist in order to grade the laryngoscopic view.
  Interventions: Procedure: Measurements of thyromental distances, hyomental distances and neck circumferences

INTERVENTIONS:
Procedure: Measurements of thyromental distances, hyomental distances and neck circumferences — thyromental distances, hyomental distances and neck circumferences using measurement tape by two independent investigators.

SUMMARY:
Difficult intubation is the situation that anesthesiologists don't want to face. Sometimes, difficult intubation affects the patient's oxygen saturation and harms for life. Many studies try to identify the predictors of difficult airway in pediatric patients. In this study, the investigator team want to identify the predictors of difficult intubation in pediatric patient by using additional parameters which are including hyomental distance, sternomental distance, neck circumference, ratio of hyomental distance to Thyromental distance, ratio of hyomental distance to sternomental distance, ratio of height to neck circumference, ratio of height to thyromental distance, Ratio of height to hyomental distance.

DETAILED DESCRIPTION:
After approval from the instution's Ethics Committee, a prospective cohort study was conducted in pediatric patients aged between 1-8 years, ASA physical status I-II who were scheduled for general anesthesia in elective surgery. One day prior surgery, Children and their parents were invited to be participated in the study by using verbal invitation and flyer. After giving consent, Addition physical examinations which are the measurements of hyomental distance, sternomental distance and neck circumference were done by two independent investigators. The ratio of hyomental distance to Thyromental distance, ratio of hyomental distance to sternomental distance, ratio of height to neck circumference, ratio of height to thyromental distance and ratio of height to hyomental distance. At the day of surgery, standard general anesthesia (balance technique) was done. The child was intubated using aged appropriated laryngoscope by general anesthesiologist. Cormack-Lehane grading was used to identify the difficult intubation. (grade III and IV). Data will be analyzed by R Program. The statistically significance was set as P<0.05. Multivariate Logistic Regression analysis will be used to identify the predictors of difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged between 1-8 years
* Schedule for elective surgery
* Having balance Anesthesia technique for surgery

Exclusion Criteria:

* Having aspiration risks
* Having history of difficult airway
* Abnormality of cervical spine /head and neck area
* Parental refusion

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged between 1-8 years who schedule for elective surgery and having balance Anesthesia technique for surgery
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
The predictors of difficult airway | up to 1 minutes after starting the process of intubation
  Laryngoscopic view was determined by using Cormack-Lehane grading (grade III-IV) were used to identify difficult intubation situation

SECONDARY OUTCOMES:
The correlation between time spent for intubation and laryngoscopic view | up to 10 minutes after starting the process of intubation
  Laryngoscopic view was determined by using Cormack-Lehane grading (grade III-IV) were used to identify difficult intubation situation

CONTACTS AND LOCATIONS:
Locations (1):
- Ngamjit Pattaravit, Songkhla, Thailand